CLINICAL TRIAL: NCT01033929
Title: A Safety and Dose Finding Trial of the Diagnostic Test C-Tb, When Given Intradermally by the Mantoux Technique to Adult Patients Recently Diagnosed With Active TB
Brief Title: A Safety and Dose Finding Trial of C-Tb, When Given to Adult Patients Recently Diagnosed With Active Tuberculosis
Acronym: TESEC-02
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Statens Serum Institut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: TESEC-02; 2009-012984-33 (Other: EudraCT Number)
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Tuberculosis
Keywords: tuberculosis; ESAT-6; CFP-10; skin test; diagnostic test
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.01µg C-Tb (Experimental): 12-24 patients depending on a safety evaluation will receive a low dose of 0.01 µg/0.1 mL C-Tb without phenol in the RIGHT or LEFT arm and 0.01 µg/0.1 mL C-Tb with phenol in the opposite arm, in a double blind manner.
  Interventions: Biological: rdESAT-6 + rCFP-10 (C-Tb)
- 0.1µg C.Tb (Experimental): 12-24 patients depending on a safety evaluation will receive a high dose of 0.1 µg/0.1 mL C-Tb without phenol in the RIGHT or LEFT arm and 0.01 µg/0.1 mL C-Tb with phenol in the opposite arm, in a double blind manner.
  Interventions: Biological: rdESAT-6 + rCFP-10 (C-Tb)

INTERVENTIONS:
Biological: rdESAT-6 + rCFP-10 (C-Tb) — rdESAT-6 + rCFP-10 (C-Tb) skin test +/- phenol administered intradermally by the mantoux injection technique. Each patient receives the unpreserved version in one arm and the preserved version in the other arm in double blind manner.
  Other Names: rdESAT-6 + rCFP-10; C-Tb

SUMMARY:
The primary objective is to assess the safety of two doses of C-Tb (0.01 and 0.1 µg/0.1 mL) when administered intradermally by the Mantoux technique to patients in the acute phase of treatment against active TB. The secondary objectives are to assess the immune response of two doses (0.01 and 0.1 µg/0.1 mL) of C-Tb from the size of induration and to assess the safety of unpreserved C-Tb and C-Tb preserved with 0.5% phenol (local reactions).

DETAILED DESCRIPTION:
This clinical trial is a single centre phase Ib open dose adjustment study with respect to the dose of C-Tb combined with a double blind randomised, split-body comparison of unpreserved C-Tb and C-Tb preserved with 0.5% phenol (each patient receives the unpreserved version in one arm and the preserved version in the other arm).

ELIGIBILITY:
Inclusion Criteria:

The patient:

1. Has signed an informed consent
2. Is willing and likely to comply with the trial procedures
3. Has been diagnosed with active TB and has been in treatment ≤ 60 days at the time of inclusion

   * has 1 documented positive sputum smear microscopy result
   * has positive culture
   * has a positive PCR result for tuberculosis
   * has a compatible clinical picture of TB with the intention to treat
4. Has a positive T-spot assay or a QuantiFERON®-TB Gold In Tube test
5. Is prepared to grant authorized persons access to their medical records

Exclusion Criteria:

The patient:

1. Has been in treatment with a product which is likely to modify the immune response within 3 months prior to the day of inclusion (e.g., immunoglobulin, systemic corticosteroids, methotrexate, azathioprine, cyclosporine or blood products)
2. Has been vaccinated with a live vaccine within 6 weeks prior to the day of inclusion (e.g. BCG, MMR, yellow fever, oral typhoid vaccines)
3. Has a known congenital or acquired immune deficiency
4. Has a disease affecting the lymphoid organs (e.g., Hodgkin's disease, lymphoma, leukaemia, sarcoidosis)
5. Is infected with HIV
6. Has severe scarring, burn, rash, eczema, psoriasis, or any other skin disease at or near the injection sites
7. Has a condition where blood drawings pose more than minimal risk for the patient, such as haemophilia, other coagulation disorders, or significantly impaired venous access
8. Is actively participating in another clinical trial
9. Is pregnant according to urine pregnancy test at inclusion
10. Has a condition which in the opinion of the investigator is not suitable for participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Local and systemic adverse reactions at the injection sites within 28 days after application of the tests (0.01/0.1 µg C-Tb). | Within 28 days after the injections

SECONDARY OUTCOMES:
Immune response of 2 doses (0.01 and 0.1 µg/0.1 mL) of C-Tb from the size of induration; the safety of unpreserved C-Tb and C-Tb preserved with 0.5% phenol and the pain associated with the injection of unpreserved C-Tb and preserved C-Tb | Within 28 days after the injections

CONTACTS AND LOCATIONS:
Overall Officials: Pernille N Tingskov, Study Director — Statens Serum Institut; David JM Lewis, Professor, Principal Investigator — St George's, University of London
Locations (1):
- St George's University of London, London, London SW17 0RE, United Kingdom

REFERENCES:
- [Derived] Aggerbeck H, Giemza R, Joshi P, Tingskov PN, Hoff ST, Boyle J, Andersen P, Lewis DJ. Randomised clinical trial investigating the specificity of a novel skin test (C-Tb) for diagnosis of M. tuberculosis infection. PLoS One. 2013 May 14;8(5):e64215. doi: 10.1371/journal.pone.0064215. Print 2013. PMID 23691171